CLINICAL TRIAL: NCT07294196
Title: Effectiveness of Percutaneous Electrolysis Treatment Targeting the Muscle-Fascia Chain in Chronic Plantar Fasciitis: A Randomized Controlled Study
Brief Title: Percutaneous Electrolysis Targeting the Muscle-Fascia Chain for Treating Chronic Plantar Fasciitis in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sivas State Hospital (Other)
Responsible Party: Principal Investigator, Serkan Polat, MD, Sivas State Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPTE-PF-001-S
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plantar Fascia Percutaneous Electrolysis plus Exercise (Active Comparator): Participants receive a conventional home-based exercise program including plantar fascia and Achilles tendon stretching, ball or roller rolling, and towel-grasping exercises targeting the intrinsic foot muscles, plus three sessions of ultrasound-guided percutaneous electrolysis applied only to the plantar fascia on days 1, 8, and 14, using 0.3-mm acupuncture needles and an EPTE® percutaneous electrolysis device (350 µA, 80 seconds).
  Interventions: Other: Exercise; Device: Percutaneous Electrolysis
- Muscle-Fascia Chain Percutaneous Electrolysis plus Exercise (Experimental): Participants receive the same conventional home-based exercise program as the active comparator group, plus three sessions of ultrasound-guided percutaneous electrolysis applied to both the plantar fascia and the myofascial trigger points of the gastrosoleus muscles on days 1, 8, and 14, using 0.3-mm acupuncture needles and an EPTE® percutaneous electrolysis device (350 µA, 80 seconds).
  Interventions: Other: Exercise; Device: Percutaneous Electrolysis

INTERVENTIONS:
Other: Exercise — Conventional home-based exercise program consisting of plantar fascia and Achilles tendon stretching, ball or roller rolling under the foot, and towel-grasping exercises targeting the intrinsic foot muscles. Participants are instructed to perform the exercises daily for the duration of the treatment period.
Device: Percutaneous Electrolysis — Ultrasound-guided percutaneous electrolysis performed with 0.3-mm acupuncture needles connected to an EPTE® percutaneous electrolysis device (Ionclinics & A. Deionic SL, Valencia, Spain). A direct galvanic current of 350 µA is applied for 80 seconds per point in each session. Three treatment sessions are administered on days 1, 8, and 14. In the active comparator arm the procedure is applied only to the plantar fascia, whereas in the experimental arm it is applied to both the plantar fascia and the myofascial trigger points of the gastrosoleus muscles.

SUMMARY:
The aim of this study is to compare, in terms of treatment effectiveness, a control group receiving a combination of a conventional exercise program and percutaneous electrolysis applied to the plantar fascia with an intervention group receiving a combination of a conventional exercise program plus percutaneous electrolysis applied both to the plantar fascia and to myofascial trigger points in the gastrosoleus muscles. Patients participating in the study will be randomized into two groups. Both groups will receive a conventional home exercise program. In the intervention group, percutaneous electrolysis treatment will be applied to both the plantar fascia and the trigger points of the gastrosoleus muscles. In the control group, percutaneous electrolysis treatment will be applied only to the plantar fascia. The percutaneous electrolysis treatment protocol will be administered on the 1st, 8th and 14th days of treatment under ultrasound guidance, using 0.3-millimeter acupuncture needles and an EPTE® percutaneous electrolysis device (Ionclinics & A. Deionic SL, Valencia, Spain) at an intensity of 350 µA for 80 seconds. The conventional home exercise program will include plantar fascia and Achilles tendon stretching, ball or cylinder rolling, and towel-grasping exercises targeting the intrinsic foot muscles. Patients' subjective pain intensity will be assessed using the Visual Analog Scale (VAS), pressure pain threshold using an algometer, functional level using the Foot Function Index (FFI), tissue parameters using ultrasound, and maximum standing and walking times without heel pain; all outcomes will be measured and recorded before treatment, after treatment, and three months after the start of treatment. The aim of the study is to compare, in terms of treatment effectiveness, the control group receiving a combination of a conventional exercise program and percutaneous electrolysis applied to the plantar fascia with the intervention group receiving a combination of a conventional exercise program plus percutaneous electrolysis applied to both the plantar fascia and the myofascial trigger points in the gastrosoleus muscles.

ELIGIBILITY:
Inclusion Criteria:

Patients who agree to participate in the study, are between 18 and 70 years of age, have had symptoms for at least 6 weeks, and have a diagnosis of plantar fasciitis confirmed clinically (sharp pain on the plantar surface of the foot upon standing after rest, heel pain that is most severe with the first steps in the morning and decreases with mild activity) and by ultrasonography (plantar fascia thickness recorded as >4 mm on ultrasound), who have not previously received any medical treatment for the condition, who agree not to use anti-inflammatory drugs during the treatment period, who have normal blood laboratory findings, who have no known acute or chronic inflammatory disease, who have a level of education sufficient to understand the treatment and procedures applied, and who are able to complete the treatment evaluation forms will be included in the study.

Exclusion Criteria:

Patients with malignancy, active infection, a history of systemic inflammatory rheumatic disease, trauma, skin lesions, infection or open wounds on the foot, neuropathy, radiculopathy, peripheral circulatory disorders, coagulopathy, warfarin use, arthropathy, congenital or acquired lower extremity deformity, sequelae of lower extremity fracture, the presence of a prosthesis, internal plate or screw fixation, a cardiac pacemaker, a metal implant in the treatment area, conditions that contraindicate physiotherapy such as pregnancy, or metal allergy will not be included in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (VAS) | Baseline (before treatment), immediately after completion of the 3rd treatment session (approximately 2 weeks), and 3 months after treatment initiation.
  Pain intensity related to plantar heel pain will be assessed using a 10-cm Visual Analog Scale (VAS). Higher scores indicate greater pain.

SECONDARY OUTCOMES:
Change in Pressure Pain Threshold (Algometry) | Baseline, post-treatment (approximately 2 weeks), and 3 months after treatment initiation.
  Pressure will be applied with an algometer at a right angle to the point on the plantar fascia where tenderness is most pronounced, and the patient will be asked to indicate the level at which discomfort is felt. The pressure value at which pain occurs will be determined as the pain threshold, and the pressure-pain threshold will be objectively assessed and recorded. Measurements will be repeated three times, and the best value will be recorded.
Change in Functional Status (Foot Function Index - FFI) | Baseline, post-treatment (approximately 2 weeks), and 3 months after treatment initiation.
  Foot-related pain and disability will be evaluated using the Foot Function Index (FFI). Higher scores indicate greater pain and functional limitation.
Change in Ultrasound Tissue Parameters of the Plantar Fascia | Baseline, post-treatment (approximately 2 weeks), and 3 months after treatment initiation.
  Tissue characteristics of the plantar fascia (e.g., thickness and echotexture, presence of hypoechogenic areas or neovascularization) will be assessed using musculoskeletal ultrasound.
Change in Maximum Pain-Free Standing and Walking Time | Baseline, post-treatment (approximately 2 weeks), and 3 months after treatment initiation.
  The maximum time that participants can stand and walk on a flat surface without plantar heel pain will be recorded using a stopwatch. Longer times indicate better functional capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Devlet Hastanesi, Sivas, Merkez, Turkey (Türkiye)